CLINICAL TRIAL: NCT01165489
Title: Discovering Laryngomalacia
Status: Completed | Type: Observational
Sponsor: Boushahri Clinic Medical Center (Other)
Responsible Party: Medical Director, Dr Mohamed Said EL-Sayed
Other Study IDs: Boushahri Medical Center
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2009-12

CONDITIONS: Laryngomalacia
Keywords: Laryngomalacia; Congenital Anomalies; Associated Health Problems
MeSH Terms: conditions — Laryngomalacia; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Laryngomalacia: Patients with Laryngomalacia
- Control Group: Patients without Laryngomalacia

SUMMARY:
Laryngomalacia is the most common congenital malformation of the larynx. It results from abnormal prolapse of supraglottic structures during inspiration. Symptoms usually appear within the first 2 weeks of life. Its severity increases in up to 6 months. 15-60% of infants with laryngeomalacia have synchronous airway anomalies.

DETAILED DESCRIPTION:
500 full term babies ≥37 weeks of both sexes delivered by different modes of delivery, with birth weights ≥2.5 kg, no history of natal or post-natal complications and from the same community. Mothers of these babies are from different socioeconomic standards and from the same community. These babies were diagnosed as having laryngomalacia. Clinical, flexible nasal and laryngeal scope, radiological and milk scintiscan were the tools used in our assessment. One thousand full term babies delivered with normal larynx, almost within the same period of time and from the same community were used as a control.

Laryngomalacia was recognized with significant statistical difference in dacryostenosis, deviated nasal septum, adenoid hypertrophy and gastroesophageal reflux disease. No significant statistical difference in pectus excavatum, cleft lip or palate, congenital lobar emphysema fistula and choanal atresia.

ELIGIBILITY:
Inclusion Criteria:

* 500 full term babies ≥ 37 weeks of both sexes were delivered by different modes of delivery, with birth weights of ≥ 2.5 kg, with no history of natal complications and from the same community.
* Mothers of these babies are from different socioeconomic standards with different educational levels.

Exclusion Criteria:

-

Ages: 4 Weeks to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S EL-Sayed, MBBCh, MSc, MD, Principal Investigator — New Children's Hospital, Cairo University
Locations (1):
- Boushahri Clinic Medical Center, Kuwait City, Kuwait